CLINICAL TRIAL: NCT05591638
Title: Comparison of Docosahexaenoic Acid Serum Levels in Patients With Preeclampsia and Control Group
Brief Title: Docosahexaenoic Acid Serum Levels in Patients With Preeclampsia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Senol Senturk, Associate professor, Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: 2022/169
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; docosahexaenoic acid; fatty acids; omega-3
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GROUP 1: There will be 45 patients diagnosed with preeclampsia in the study group
- GROUP 2: There will be 45 normal pregnant women in the control group

SUMMARY:
By comparing the blood levels of docosahexaenoic acid (DHA) in preeclamptic patients with normal pregnant women, we aim to reveal the relationship between these markers, which are known to be effective on metabolic function, and preeclampsia, and to contribute to future studies and possible treatment options

DETAILED DESCRIPTION:
The research is a prospective cross-sectional study to be conducted at Recep Tayyip Erdogan University Training and Research Hospital, Department of Obstetrics and Gynecology. The current treatments of the patients will not be changed and no medical treatment or interventional procedures will be applied to the patients for study purposes. After the patients are informed about the study, the consent form will be signed, indicating that they voluntarily participated in the study. Apart from the biochemical parameters required for the diagnosis and treatment of the patients, different parameters will not be considered. The supply of Docosahexaenoic Acid kits required for the study will be provided by the executive physician and the blood taken from the patients will be evaluated.

G * Power 3.1.9.7 program was used to calculate the sample size for this study. At 80% statistical power and α=0.05 significance level, the smallest required sample size was calculated as 86 (control 44- study: 42) when d=0.51 effect size was calculated according to t-test for independent groups. Considering that there may be missing data, 90 patients between the ages of 18-40 will be included in the study. There will be 45 patients diagnosed with preeclampsia in the study group. There will be 45 normal pregnant women in the control group.

Preeclamptic patient selection and classification will be made according to the 2019 diagnostic criteria of the American Society of Obstetrics and Gynecology (ACOG). Accordingly, the diagnosis of preeclampsia; After 20 weeks of gestation in a normotensive pregnant woman, hypertension (systolic ≥140 mmHg and/or diastolic ≥90 mmHg) proteinuria or thrombocytopenia with hypertension (platelet <100,000/103 /μL), impaired liver function tests (liver liver function) transaminase blood values to twice the normal concentration), new-onset renal failure (serum creatinine values > 1.1 mg/dL or a two-fold increase in serum creatinine in the absence of other renal disease), pulmonary edema, or new-onset cerebral and visual acuity will be placed in case of malfunctions. proteinuria; Proteinuria ≥ 300 mg in 24-hour urine or protein/creatinine ratio ≥ 0.3 or 1+ proteinuria as measured by urine stick. The diagnosis of severe preeclampsia will be made when blood pressure values are systolic ≥160 mmHg and/or diastolic ≥110 mmHg.

Demographic, clinical and laboratory data of the pregnant women included in the study will be recorded. The last menstrual period, obstetric examination and ultrasonography findings will be taken as basis in the determination of the gestational week. For each patient, age, body mass index (BMI), number of births, week of birth, type of birth, birth weight, complete blood count (hemogram), liver function tests (AST, ALT), kidney function tests (urea, creatinine) and full Urine test results will be recorded. In order to avoid the possible effects of corticosteroid and MgSO4 treatments on laboratory parameters in preeclamptic pregnant women, the first laboratory results at hospitalization will be taken into account. In addition, 1st and 5th minute APGAR scores will be noted to assess perinatal outcomes.

Inclusion criteria: Pregnant women aged 18-40, singleton pregnancies, pregnant women with preeclampsia, healthy pregnant women without a history of hypertension before and after pregnancy

Exclusion criteria:

Pregnant women diagnosed with chronic hypertension before pregnancy, pregnant women with hypertension before the 20th gestational week, multiple pregnancies, pregnant women with molar pregnancies, women with a body mass index (BMI) >30kg/m2, pregnant women with a history of birth complicated with chromosomal abnormalities, pre-pregnancy or during pregnancy Pregnant women diagnosed with diabetes mellitus, pregnant women diagnosed with chronic systemic diseases, especially rheumatological, renal and vascular diseases, pregnant women diagnosed with chorioamnionitis, pregnant women with polyhydramnios, maternal infection diagnosis.

In the study, since the medical treatment of the patients was not changed and additional medical treatment and interventional procedures were not applied, it would not be necessary to take safety precautions. The blood taken from the patients for routine diagnosis and treatment will be stored at -20 degrees Celsius after the serum and plasma are separated. By comparing the blood levels of docosahexaenoic acid (DHA) in preeclamptic patients with normal pregnant women, the relationship between these markers, which are known to be effective on metabolic function, and preeclampsia will be evaluated. Afterwards, follow-up, treatment and laboratory evaluation for study purposes are not required.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the ages of 18-40, singleton pregnancies, pregnant women with preeclampsia, healthy pregnant women who do not have a history of hypertension before and after pregnancy

Exclusion Criteria:

* Pregnant women diagnosed with chronic hypertension before pregnancy, pregnant women with hypertension before the 20th gestational week, multiple pregnancies, pregnant women with molar pregnancies, women with a body mass index (BMI) >30kg/m2, pregnant women with a history of birth complicated with chromosomal abnormalities, pre-pregnancy or during pregnancy Pregnant women diagnosed with diabetes mellitus, pregnant women diagnosed with chronic systemic diseases, especially rheumatological, renal and vascular diseases, pregnant women diagnosed with chorioamnionitis, pregnant women with polyhydramnios, maternal infection diagnosis

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: 18-40 years old pregnant women at 20-40 weeks of gestation with and without preeclampsia (study and control)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-10-24 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
docosahexaenoic acid | 6 months
  docosahexaenoic acid levels between groups will be measured

CONTACTS AND LOCATIONS:
Overall Officials: SENOL SENTURK, Study Director — Recep Tayyip Erdogan University

IPD SHARING:
Plan to Share IPD: Undecided